CLINICAL TRIAL: NCT06359743
Title: Ultrasound Guided Quadratus Lumborum Block Versus Laparoscopic Superior Hypogastric Plexus Block for Postoperative Analgesia After Laparoscopic Hysterectomy
Brief Title: Ultrasound Guided QLB Versus Laparoscopic Superior Hypogastric Plexus Block for Postoperative Analgesia After Laparoscopic Hysterectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Abdalla Mohamed Goda Mohamed, Abdalla mohamed goda mohamed ,MD, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 271/7
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Post Hysterectomy Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group QL: (Experimental): patients will receive Ultrasound Guided bilateral QL lumborum block (Anterior Approch) by anesthesiologist (20 ml of 0.25% bupivacaine hydrochloride at each side).
  Interventions: Procedure: Quadratus Lamborum versus superior hypogatric
- Group SH: (Experimental): will receive laparoscopic Superior Hypogastric block by gynecologist (30 ml of 0.25% bupivacaine hydrochloride ).
  Interventions: Procedure: Quadratus Lamborum versus superior hypogatric

INTERVENTIONS:
Procedure: Quadratus Lamborum versus superior hypogatric — Ultrasound Guided Quadratus Lumborum Block versus Laparoscopic Superior Hypogastric Plexus Block for Postoperative Analgesia after Laparoscopic Hysterectomy

SUMMARY:
Pain following laparoscopic hysterectomy may interfere with early ambulation, discharge of patient from hospital and interfere with enhanced recovery with more opioid consumption. Most of methods for postoperative pain depend on the use of high doses of opioids with more side effects such as nausea, vomiting, respiratory center depression, delay bowel motility and hemodynamics instability. To decrease of opioid consumption in postoperative pain management as well as related side effects, previous studies showed that quadratus lumborum block or superior hypogastric plexus block (SHPB) had shown promising success in management of postoperative pain in patients undergoing laparoscopic hysterectomy. The present study will be conducted to compare of ultrasound guided QL block and laparoscopic superior hypogastric plexus block as a part of multimodal analgesia may allow adequate analgesia and decrease the overall use of opioids and allow patient enhanced recovery.

DETAILED DESCRIPTION:
hypothesis: There is no difference between the analgesic effect of either Ultrasound guided QL block or laparoscopic Superior hypogastric plexus block on post laparoscopic hysterectomy pain.

Alternative hypothesis:

There is difference between the analgesic effect of either Ultrasound QL block or laparoscopic superior hypogastric plexus block on post laparoscopic hysterectomy pain.

Aim of the work Better achievement of effective analgesia with less opioid consumption and related side effects for post laparoscopic hysterectomy pain.

Objectives To assess effect of both ultrasound quadratus lumborum block and laparoscopic superior hypogastric plexus block on analgesic outcome (Visual Analogue Scale VAS, duration of analgesia) after laparoscopic hysterectomy. To compare between ultrasound quadratus lumborum block and laparoscopic superior hypogastric plexus block regarding to total opioid for postoperative analgesia after laparoscopic hysterectomy and patient satisfaction. To record side effects related to regional block ( e.g., local anesthetic toxicity, vascular and neural injury) and opioids ( neasuea, vomiting, respiratory depression

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from the patient.
2. BMI of less than or equal 30.0 kg m-2.
3. Age 45-60 years old.
4. American Society of Anesthesiologists (ASA) physical status classes I and II.Exclusion Criteria:

1. Allergy to local anesthetics. 2. Infection at site of injection. 3. Patients with coagulopathy. 4. Patients with chronic pain syndromes. 5. Physical and mental disease which could interfere with pain scores evaluation.

6. Patients with distorted local anatomy.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption decrease | 24hours
  Avoid excessive usage of opioid by regional blocks

CONTACTS AND LOCATIONS:
Overall Officials: Eslam S Almaghawry Mohamed, MD, Study Chair — Faculty of medicine, Zagazig university; Abdalla H Gad, MD, Study Chair — Faculty of medicine, zagazig university; Mohamed A Wasfy, MD, Study Chair — Faculty of medicine, zagazig university
Locations (1):
- Faculty of medicine, Zagazig university, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Blanton E, Lamvu G, Patanwala I, Barron KI, Witzeman K, Tu FF, As-Sanie S. Non-opioid pain management in benign minimally invasive hysterectomy: A systematic review. Am J Obstet Gynecol. 2017 Jun;216(6):557-567. doi: 10.1016/j.ajog.2016.12.175. Epub 2016 Dec 30. PMID 28043841
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233